CLINICAL TRIAL: NCT07296081
Title: Myocardial Fibrosis in Heart Failure: A Pilot Study With 68Ga-FAPI PET/CT
Brief Title: ⁶⁸Ga-FAPI PET/CT for Cardiac Fibrosis in Heart Failure
Acronym: MY-FAPI
Status: Recruiting | Type: Observational
Sponsor: University of Coimbra (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, João Pedro Borges Rosa, MD, Cardiologist, PhD Student, University of Coimbra
Other Study IDs: CE-113/2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Fibrosis; Heart Failure
Keywords: Fibroblast activation protein inhibitors; Gallium-68; Heart failure; Myocardial fibrosis; Positron emission tomography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with HFrEF and HFpEF: patients with HFrEF (non-ischemic dilated cardiomyopathy) and HFpEF (hypertrophic cardiomyopathy)
  Interventions: Diagnostic Test: 68Ga-FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/CT — Positron emission tomography/computed tomography (68Ga-FAPI PET/CT)

SUMMARY:
Heart failure (HF) is a clinical syndrome with increasing incidence and prevalence, associated with high morbidity, mortality, and economic impact, despite therapeutic advances.

Myocardial fibrosis is a common feature across different pathophysiological processes and plays a key role in HF development, with growing research interest specifically in non-ischemic dilated cardiomyopathy (HFrEF phenotype) and hypertrophic cardiomyopathy (HFpEF phenotype). Given its potential reversibility with certain drugs, fibrosis is an attractive therapeutic target, requiring non-invasive methods to monitor fibrogenesis and treatment efficacy.

Cardiac magnetic resonance imaging (CMR) is the gold standard for detecting fibrosis but cannot distinguish between active and inactive fibrosis or detect early stages, limitations that may be addressed by gallium-68-labeled fibroblast activation protein inhibitor positron emission tomography/computed tomography (68Ga-FAPI PET/CT).

This single-center, prospective, observational pilot study aims primarily to assess myocardial fibrosis in patients with HFrEF (non-ischemic dilated cardiomyopathy) and a subtype of HFpEF (hypertrophic cardiomyopathy) using 68Ga-FAPI PET/CT compared to CMR.

Secondary objectives include developing 68Ga-FAPI uptake assessment methodologies for future anti-fibrotic therapy studies and correlating fibrosis with serum cardiac biomarkers and cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Signs and symptoms of heart failure (HF);
* [Preserved left ventricular ejection fraction (LVEF) (≥50%) and Evidence of structural/functional abnormality consistent with diastolic dysfunction/increased ventricular filling pressures, including elevated natriuretic peptides and Imaging diagnosis of hypertrophic cardiomyopathy and Genetic diagnosis of hypertrophic cardiomyopathy due to sarcomeric gene mutation] OR [Reduced LVEF (≤40%) and Imaging diagnosis of dilated cardiomyopathy: left ventricular end-diastolic diameter >58 mm in men and >52 mm in women, and left ventricular volume ≥75 mL/m² in men and ≥62 mL/m² in women, not explained solely by loading conditions]
* Recent transthoracic echocardiogram (< 3 months);
* Recent cardiac magnetic resonance imaging (< 3 months).
* Normal coronary angiogram or computed tomography coronary angiography within 6 months of enrolment

Exclusion Criteria:

* Inability to provide informed consent;
* Inability to tolerate the supine position;
* Hemodynamic instability;
* Claustrophobia;
* Chronic kidney disease with glomerular filtration rate <30 mL/min/1.73m²;
* Pregnant or breastfeeding women;
* Malignant neoplasms within the past 5 years;
* Significant primary valvular disease;
* Significant atherosclerotic coronary artery disease;
* Grade 2 or 3 arterial hypertension;
* Presence of an implanted cardiac electrical device;
* Recent hospitalization for heart failure (<30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen patients with HFrEF (non-ischemic dilated cardiomyopathy) and Fifteen patients with HFpEF (hypertrophic cardiomyopathy)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
68Ga-FAPI uptake | Baseline
  Comparison of myocardial fibroblast activation identified by 68Ga-FAPI PET/CT with the non-invasive gold standard for fibrosis detection (Cardiac magnetic resonance with late gadolinium enhancement and extracellular volume)

SECONDARY OUTCOMES:
68Ga-FAPI uptake | Baseline (1 & 2) and after 2 years (3)
  1. Identify suitable methodologies for assessing 68Ga-FAPI uptake for future studies evaluating the efficacy of anti-fibrotic therapies.
  2. Correlate myocardial fibroblast activation identified by 68Ga-FAPI PET/CT with serum markers of cardiac pathology.
  3. Correlate myocardial fibroblast activation identified by 68Ga-FAPI PET/CT with cardiovascular events over a 2-year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade de Coimbra, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided